CLINICAL TRIAL: NCT00984594
Title: Evaluation of the Composite of Cancellous and Demineralized Bone Plug (CR-Plug) for Repair of Osteochondral Defects in High-Load-Bearing Region and Low-Load-Bearing Region of the Femoral Condyle
Brief Title: Evaluation of a Composite Cancellous and Demineralized Bone Plug (CR-Plug) for Repair of Knee Osteochondral Defects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrolment & potential regulatory changes for allograft in cartilage repair
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR2008
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Knee Injury
Keywords: allograft; knee injury; cartilage injury
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary injury site (Other): CR-Plug will be placed in the site of the primary injury
  Interventions: Other: Primary injury site
- Backfill site (Other): Autograft will be placed in the site of the primary injury; CR Plug will be placed in the harvest site
  Interventions: Other: Backfill site

INTERVENTIONS:
Other: Primary injury site — Autograft will be placed in the primary defect site.
  Arms: Primary injury site
Other: Backfill site — Autograft will be placed in the primary defect site; CR-Plug will be placed in the harvest site.
  Arms: Backfill site

SUMMARY:
The objective of this study is to determine how effective a plug made out of human bone (called "CR-Plug") will be in the treatment of smaller, focal defects (like the injury the patient has to their knee).

DETAILED DESCRIPTION:
The main objective of this double arm study is to test the ability of an allograft plug to provide "successful" repair of less than (<) 2.5 cm2 osteochondral defect in a low-load-bearing femoral condyle region, and a high-load-bearing femoral-condyle region.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years
* skeletally mature
* Have a symptomatic score International Cartilage Repair Society (ICRS) grade 3a, 3b, 3c, 3d, 4a, 4b articular cartilage lesion less than 2.5 cm involving the Medial Femoral Condyle or Lateral Femoral Condyle. Symptoms must include pain, pain with weight bearing and squatting, locking of joints and or swelling
* Functional meniscal tissue (defined as 5 mmor greater)
* A score of = or greater than 4 on the VAS questionnaire

Exclusion Criteria:

* Associated tibial or patellar articular cartilage defect greater than 2 ICRS
* Osteoarthritis of either knee
* Mechanical axis malalignment of greater than 5 degrees
* Patellofemoral incongruity on Merchant view
* One or more multiple defects greater than 2.5 cm
* Osteochondritis dissecans (OCD) with depth of bone loss greater than 4 mm
* Ligament treatments in the affected knee within one year prior to current study
* Previous surgical meniscus treatment in the affected knee in the last 6 months
* Less than 5 mm of meniscal tissue in ipsilateral compartment of study treatment
* use of any investigational therapy within 30 days prior to the first visit
* Corticosteroid or viscosupplementation within the past 3 months
* A score of 3 or less on the VAS questionnaire
* Active gout or pseudogout or systemic inflammatory condition
* Microfracture less than one year prior to current study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akbar Nawab, MD, Principal Investigator — Ellis and Badenhausen Orthopaedics, PSC
Locations (1):
- Ellis and Badenhausen Orthopaedics, PSC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the patient population at one of the investigative sites between 12 June 2009 and 5 May 2010.
  One subject was enrolled at 17 years, 7 months. A protocol waiver was approved by the Institutional Review Board and parental informed consent and assent of subject was obtained.
Pre-assignment Details: Patients were assigned to the treatment arm based on a randomization table. Enrolled patients excluded: Not fulfilling inclusion or exclusion criteria, withdrawal of consent. Enrolled patients were followed to completion unless lost to follow up. Of 4 enrolled, 1 withdrew consent, 1 was lost to follow up & 2 completed
Groups:
- Backfill: Autograft will be placed in the primary defect site, CR Plug will be placed in the harvest site.
- Primary: CR Plug will be placed in the site of the primary injury.
Period: Overall Study
Arm/Group | Backfill | Primary
Started | 2 | 2 (One patient withdrew consent and left the study before treatment.)
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: There are only 3 patients in the baseline analysis due to one patient withdrawing from the study before data collection.
Groups:
- Backfill: Autograft will be placed in the primary defect site; CR Plug will be placed in the harvest site
- Total: Total of all reporting groups
Arm/Group | Backfill | Primary | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (12.02) | 17 (0) | 24.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS
Description: The outcome at 24 months as measured by the Knee injury and Osteoarthritis Outcome Score (KOOS). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Time Frame: 24 months
Population: Of the 2 patients enrolled in the backfill group, 1 was lost to follow-up, therefore the data presented is for only 1 patient.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Backfill | Primary
Number analyzed (Participants) | 1 | 1
units on a scale | 82.74 [82.74 to 82.74] | 100 [100 to 100]

2. Secondary Outcome: Current Health Assessment (CHA)
Description: Evaluation on the Current Health Assessment at 24 months. Scores are transformed to a 0-100 scale, with zero representing a self-graded perception of extremely poor health and 100 representing no health problems. Scores between 0 and 100 represent the percentage of total possible score achieved.
Time Frame: 24 months
Population: Of the 2 patients enrolled in the study in the backfill group, 1 was lost to follow-up, therefore the data presented is for only 1 patient.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Backfill | Primary
Number analyzed (Participants) | 1 | 1
units on a scale | 80.6 [80.6 to 80.6] | 100 [100 to 100]

3. Secondary Outcome: IKDC Assessment
Description: The International Knee Documentation Committee (IKDC) scores from 24 months are shown. The IKDC is an index score from 0 to 100, with 100 being the best possible score,
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Backfill | Primary
Number analyzed (Participants) | 1 | 1
units on a scale | 74.7 [74.7 to 74.7] | 98.6 [98.6 to 98.6]

4. Secondary Outcome: Magnetic Resonance Imaging (MRI) Results
Description: MRI images were graded by a radiologist with regard to the incorporation of the CR graft in both the cancellous and cortical portions of the bone at the graft site. The raw scores were converted to an index scale form 0 to 100, with 0 representing failure of the graft to incorporate and 100 representing complete incorporation of the graft.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Backfill | Primary
Number analyzed (Participants) | 1 | 1
units on a scale | 97.1 [97.1 to 97.1] | 100 [100 to 100]

5. Secondary Outcome: Lysholm Score at 24 Months
Description: The Lysholm scores from the 24-month exams are shown. The Lysholm score is an indexed score of knee functional ability, with 0 being the worst score and 100 being the best score, indicating no limitations in activity/function.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Backfill | Primary
Number analyzed (Participants) | 1 | 1
units on a scale | 81 [81 to 81] | 100 [100 to 100]

ADVERSE EVENTS:
Time Frame: Patients were followed through the termination of the study, i.e. 24 months
Groups:
- Backfill: CR-Plug will be placed in harvest site.
- Primary: Autograft will be placed in primary defect site.
Arm/Group | Backfill | Primary
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Backfill (N=2) | Primary (N=1)
Increased pain in right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased swelling in right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Open Reduction Internal Fixation of talus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was closed early due to slow enrollment & a potential change in the regulatory pathway for the allograft used in cartilage repair.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days